CLINICAL TRIAL: NCT04761393
Title: Characterizing Mmp12 In Sputum And Its Relationship To Emphysema And Inflammatory Endotypes
Brief Title: Characterizing Matrix Metalloproteinase-12 (MMP12) in Sputum
Status: Recruiting | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: Foresee Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: FIRH_Xe007
Record Dates: First submitted 2021-02-11; First posted 2021-02-18 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Emphysema
MeSH Terms: conditions — Emphysema | interventions — Xenon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Sputum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with emphysema and eosinophilia in blood and sputum: blood eosinophils ≥300 cells/μL and sputum eosinophils >3%
  Interventions: Procedure: Hyperpolarized 129Xe (Xenon) diffusion-weighted MRI
- Patients with emphysema and paucicellular inflammation: sputum neutrophils <65% and eosinophils <3%
  Interventions: Procedure: Hyperpolarized 129Xe (Xenon) diffusion-weighted MRI
- Patients with emphysema and sputum neutrophilia: sputum neutrophils >65% and sputum eosinophils < 3%
  Interventions: Procedure: Hyperpolarized 129Xe (Xenon) diffusion-weighted MRI

INTERVENTIONS:
Procedure: Hyperpolarized 129Xe (Xenon) diffusion-weighted MRI — Participants will inhale a one litre gas mixture containing hyperpolarized 129Xe mixed with nitrogen (N2) or helium (4He) from a one litre dose bag. Breath-hold will be up to 16 seconds

SUMMARY:
The hypothesis is that in patients with emphysema, a high MMP12 sputum and/or blood level correlates with airspace enlargement and with increased sputum Th2 immune biomarkers.

DETAILED DESCRIPTION:
Since MMP-12 apparently has a preponderant role in the genesis of emphysema and probably in airspace enlargement, its inhibition may result in an interesting targeting point in view to find specific therapies in obstructive diseases. There is abundant evidence in animal models that shows how MMP-12 blockade inhibits the development of emphysema and airway remodeling. Unfortunately, the results have not been conclusive in human models.

In the last years, pulmonary imaging biomarkers that measure airspace enlargement have been developed. In particular, the apparent diffusion coefficient (ADC), quantified by inhaled hyperpolarized gas MRI, reflects alveolar airspace size. ADC provides information consistent with histopathological findings that may be used to estimate lung disease progression and treatment response.

ELIGIBILITY:
Inclusion Criteria (COPD):

* ≥40 years of age
* Current or ex-smokers with a >10 pack year smoking history
* Have a post-bronchodilator forced expired volume in 1 second (FEV1)/forced expired vital capacity (FVC) ratio of <70% and a post-bronchodilator FEV1 value from ≥30% predicted (GOLD 1, 2 and 3), (Global Initiative for Obstructive Lung disease)
* Have a radiologist confirmed pulmonary emphysema diagnosis based on CT

Inclusion criteria for normal controls:

* No clinically significant medical condition or a history of asthma, COPD, cystic fibrosis, or other significant respiratory disorder including significant occupational or environmental exposures with ongoing respiratory symptoms.
* No current or past smoking history
* Have a post-bronchodilator FEV1/FVC ratio of >70%

Exclusion Criteria:

Any potential subject who meets any of the following criteria will be excluded from participating in the study:

* Patients with other non-COPD airway diseases
* Patients with very severe COPD (FEV1<30% predicted)
* Patients with an intercurrent exacerbation
* Patients with life expectancy less than 3 months
* Pregnant or breastfeeding
* Undergoing immunomodulatory or biologic treatment
* Use of systemic steroids in the last month
* Hospitalization in the last 12 months due to exacerbation
* Known cardiovascular comorbidity under treatment or with hospitalizations of this cause in the last year
* That they cannot perform spirometry
* Active malignancy
* Realization of lung surgery during the study period
* History of alcohol and drug abuse that prevents compliance with follow-up
* History of bronchial thermoplasty
* Participating in another study concomitantly
* MRI Related: patients who have implanted mechanically, electrically or magnetically activated device or any metal in their body which cannot be removed, including but not limited to pacemakers, artificial limb, metallic fragments of foreign body, shunt, surgical staples (including clips or metallic sutures and/or ear implants).

Ages: 40 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This is a cross-sectional study in healthy controls and patients with pulmonary emphysema.
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-11-29 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Blood and sputum matrix metalloproteinase-12 (MMP12) levels | Baseline
  Measure sputum and blood MMP12 levels
Quantify their alveolar destruction using Computed Tomography (CT) and magnetic resonance imaging (MRI) | Baseline
  The relative area of the Computed Tomography (CT) attenuation histogram with attenuation of 950 HU or less (RA950) and the 15th percentile of the CT attenuation histogram (HU15) will be generated to quantify emphysema.
  For analysis of 129Xe diffusion-weighted MR images we will employ the same approach as described by Kirby and colleagues to quantify the apparent diffusion coefficient (ADC) and generate ADC maps12 to assess airspace size.
Measure other T2 activity biomarkers in sputum | Baseline
  Sputum: enumeration of Free eosinophils granules (FEG) by none, few moderate and many
Measure other T2 activity biomarkers in sputum supernatant | Baseline
  Sputum supernatant: Levels of (interleukin) IL-4, IL-5 and IL-13, eosinophil peroxidase, transforming growth factor (TGF)-beta, Phospho-Smad2 and Phospho-Smad3 (SMAD=Small Mothers Against Decapentaplegic gene)
Measure other T2 activity biomarkers in blood | Baseline
  Ferritin in microgram per litre (ug/L)
Measure other T2 activity biomarkers in blood | Baseline
  C reactive protein (CRP) in milligram/litre (mg/L)
Compare type-2 (T2) activity biomarkers with healthy individuals in sputum | Baseline
  Sputum: enumeration of Free eosinophils granules (FEG) as few, moderate and many.
Compare type-2 (T2) activity biomarkers with healthy individuals in blood | Baseline
  Ferritin in microgram per litre (ug/L)
Compare type-2 (T2) activity biomarkers with healthy individuals in blood | Baseline
  C reactive protein (CRP) in milligram/litre (mg/L)
Compare type-2 (T2) activity biomarkers with healthy individuals in sputum supernatant | Baseline
  Sputum supernatant: Levels of IL-4, IL-5 and IL-13, eosinophil peroxidase, TGF-beta, Phospho-Smad2 and Phospho-Smad3.

CONTACTS AND LOCATIONS:
Locations (1):
- Firestone Institute for Respiratory Health, St. Joseph's Healthcare, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Shukla Y, Wheatley A, Kirby M, Svenningsen S, Farag A, Santyr GE, Paterson NA, McCormack DG, Parraga G. Hyperpolarized 129Xe magnetic resonance imaging: tolerability in healthy volunteers and subjects with pulmonary disease. Acad Radiol. 2012 Aug;19(8):941-51. doi: 10.1016/j.acra.2012.03.018. Epub 2012 May 15. PMID 22591724
- [Background] Ostridge K, Williams N, Kim V, Bennett M, Harden S, Welch L, Bourne S, Coombs NA, Elkington PT, Staples KJ, Wilkinson TM. Relationship between pulmonary matrix metalloproteinases and quantitative CT markers of small airways disease and emphysema in COPD. Thorax. 2016 Feb;71(2):126-32. doi: 10.1136/thoraxjnl-2015-207428. Epub 2015 Dec 8. PMID 26645414
- [Background] Nair P, Ochkur SI, Protheroe C, Radford K, Efthimiadis A, Lee NA, Lee JJ. Eosinophil peroxidase in sputum represents a unique biomarker of airway eosinophilia. Allergy. 2013 Sep;68(9):1177-84. doi: 10.1111/all.12206. Epub 2013 Aug 9. PMID 23931643